CLINICAL TRIAL: NCT02708238
Title: Efficacy of a Standardized Extract of Matricariae Chamomilla L., Melissa Officinalis L. and Tyndallized Lactobacillus Acidophilus (H122) Compared With Lactobacillus Reuteri (DSM 17938) and With Simethicone for the Treatment of Infantile Colic
Brief Title: Efficacy of Matricariae Chamomilla L., Melissa Officinalis L. and Tyndallized Lactobacillus Acidophilus (H122) for Infantile Colics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Erasmo Miele, Researcher, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04032016
Record Dates: First submitted 2016-03-04; First posted 2016-03-15 (Estimated); Results first posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-06

CONDITIONS: Infantile Colics
Keywords: Infantile colics
MeSH Terms: interventions — Simethicone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): All enrolled infants randomized to Group A will receive a standardized extract of Chamomilla L., Melissa Officinalis L. and tyndallized Lactobacillus Acidophilus (H122), administered at the dose of 1 ml twice a day of a commercially available solution
  Interventions: Dietary Supplement: Standardized extract of Chamomilla L., Melissa Officinalis L. and tyndallized L. Acidophilus (H122)
- Group B (Active Comparator): All enrolled infants randomized to Group B will receive Lactobacillus reuteri DSM 17938 administered at the dose of 108 colony-forming units (CFU)/day in 5 drops of a commercially available oil suspension
  Interventions: Dietary Supplement: Lactobacillus reuteri DSM 17938 (108 CFU)
- Group C (Active Comparator): All enrolled infants randomized to Group C will receive simethicone, given at a dose of 60 mg in 15 drops two times per day of a commercially available solution
  Interventions: Drug: Simethicone

INTERVENTIONS:
Dietary Supplement: Standardized extract of Chamomilla L., Melissa Officinalis L. and tyndallized L. Acidophilus (H122)
  Arms: Group A
Dietary Supplement: Lactobacillus reuteri DSM 17938 (108 CFU)
  Arms: Group B
Drug: Simethicone
  Arms: Group C

SUMMARY:
A multicenter prospective, randomized comparative study will be conducted in infants with colic, according to Rome III criteria. Enrolled infants will be assigned at random to receive Chamomilla L., Melissa Officinalis L. and tyndallized L. Acidophilus (H122), L reuteri DSM 17938 (108 CFU) or simethicone. Treatment will be given to subjects for 28 days and they will be followed for 4 weeks. Treatment success will be assessed at the end of study period. Daily crying and fussing times will be recorded in a structured diary, and maternal questionnaires will be completed to monitor changes in infant colic symptoms and adverse events.

DETAILED DESCRIPTION:
This will be a prospective, multicentre, open label, randomized, controlled trial. All consecutive infants diagnosed with IC, according to Rome III criteria, will be prospectively enrolled in a 12 months period by 3 different Pediatric Gastroenterology units: Department of Translational Medical Science, Section of Pediatrics, University of Naples "Federico II"; Institute of Pediatrics of the University of Foggia; Endoscopy and Gastroenterology Unit, Department of Pediatrics, University of Messina.

After the enrollment, all children will be randomly assigned to receive Chamomilla L., Melissa Officinalis L. and tyndallized L. Acidophilus (H122) (Group A), L reuteri DSM 17938 (108 CFU) (Group B) or Simethicone (Group C). Treatment will be given to subjects for 28 days. The study's primary outcome is defined as a reduction in the duration of average crying times, from baseline (day 0) to end of treatment (day 28). The secondary outcome measure is the number of participants who respond to treatment on days 28. Infants who experience a decrease in the daily average crying time of 50% from baseline will be considered as responders to the treatment. Parents will be instructed to complete a structured 28-day maternal diary, modified from Barr et al. in order to record the frequency of colic episodes and the daily crying and fussing time (in minutes), feeding schedule, stool frequency and characteristics, and any adverse events experienced (14). Follow-up visits will be conducted on study days 7, 14, 21 and 28 by the same study investigator. At that visit, diaries and unused study products will be returned.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of IC according to Rome III criteria (2);
2. age ≥2 weeks to 4 months;
3. breast-fed or fomula-fed infants;
4. term delivery (≥37 weeks gestation at birth);
5. 5-minute Apgar score ≥7; and 6) birth weight ≥2500 g

Exclusion Criteria:

1. a major medical problem or acute illness;
2. family history of atopy;
3. history of antibiotic treatment before or during the study;
4. history of probiotic supplementation.

Ages: 14 Days to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Staiano, Prof., Principal Investigator — Federico II University

IPD SHARING:
Plan to Share IPD: Yes
Publication

REFERENCES:
- [Derived] Martinelli M, Ummarino D, Giugliano FP, Sciorio E, Tortora C, Bruzzese D, De Giovanni D, Rutigliano I, Valenti S, Romano C, Campanozzi A, Miele E, Staiano A. Efficacy of a standardized extract of Matricariae chamomilla L., Melissa officinalis L. and tyndallized Lactobacillus acidophilus (HA122) in infantile colic: An open randomized controlled trial. Neurogastroenterol Motil. 2017 Dec;29(12). doi: 10.1111/nmo.13145. Epub 2017 Jun 30. PMID 28665038

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: All enrolled infants randomized to Group A will receive a standardized extract of Chamomilla L., Melissa Officinalis L. and tyndallized Lactobacillus Acidophilus (H122), administered at the dose of 1 ml twice a day of a commercially available solution
  Standardized extract of Chamomilla L., Melissa Officinalis L. and tyndallized L. Acidophilus (H122)
- Group B: All enrolled infants randomized to Group B will receive Lactobacillus reuteri DSM 17938 administered at the dose of 108 colony-forming units (CFU)/day in 5 drops of a commercially available oil suspension
  Lactobacillus reuteri DSM 17938 (108 CFU)
- Group C: All enrolled infants randomized to Group C will receive simethicone, given at a dose of 60 mg in 20 drops four times per day of a commercially available solution
  Simethicone
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 60 | 60 | 60
Completed | 60 | 59 | 57
Not Completed | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 60 | 59 | 57 | 176
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 60 | 59 | 57 | 176
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: Days] | 38 [14 to 86] | 35 [14 to 85] | 30 [14 to 62] | 35 [14 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 21 | 39 | 91
  Male | 29 | 38 | 18 | 85
Region of Enrollment [Number; unit: participants]
  Italy | 60 | 59 | 57 | 176

OUTCOME MEASURES:

1. Primary Outcome: Median Daily Crying Time at the End of the Treatment
Description: Median daily crying at the end of treatment (day 28).
Time Frame: 28 days of treatment
Measure: Median (Full Range); unit: minutes
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 60 | 59 | 57
minutes | 50 [30 to 180] | 55 [30 to 180] | 80 [30 to 270]

2. Secondary Outcome: Number of Responders
Description: Number of responders defined as the number of patients who experienced a decrease in the daily average crying time of 50% from baseline
Time Frame: 28 days of treatment
Measure: Number; unit: number of responders
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 60 | 59 | 57
number of responders | 57 | 47 | 38

ADVERSE EVENTS:
Arm/Group | Group A | Group B | Group C
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/59 | 0/57
Other Adverse Events (participants affected / at risk) | 0/60 | 0/59 | 0/57

LIMITATIONS AND CAVEATS:
The absence of a placebo group and the open label design represent the main limitations of this study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No